CLINICAL TRIAL: NCT00731432
Title: The Effect Of A Transmucosal Herbal Periodontal Patch (THPP) on Gingival Inflammation in Diabetic Patients
Brief Title: Herbal Periodontal Patch (THPP) for Gingival Inflammation in Diabetics
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: Izun Pharma Ltd (Industry)
Responsible Party: Dr. Y. Caine, Herzog Hospital, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-3
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2008-08

CONDITIONS: Gingival Inflammation in Diabetic Patients
Keywords: gingivitis, diabetes mellitus, herbal, oral inflammation
MeSH Terms: conditions — Gingivitis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Transmucosal Herbal Periodontal Patch (THPP)
  Interventions: Drug: Transmucosal Herbal Periodontal Patch (THPP)
- B (Placebo Comparator): Placebo Patch
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Transmucosal Herbal Periodontal Patch (THPP) — Patch applied to oral gingiva
  Other Names: Day 1: 1 patch X 3/d; Day 2-3: 1 patch X1/d; Days 4-5: no patch
  Arms: A
Drug: Placebo Patch — Identical in shape and texture to treatment patch
  Other Names: Day 1: 1 patch X 3/d; Day 2-3: 1 patch X1/d; Days 4-5: no patch
  Arms: B

SUMMARY:
Diabetes increases the incidence and severity of periodontal inflammation and disease, and periodontal disease causes an increase in the severity of diabetes by worsening glycemic control and increasing insulin resistance.The Transmucosal Herbal Periodontal Patch (THPP) is a transmucosal patch containing an herbal compound that has an anti-inflammatory effect on gingival tissue.The primary objective of this study is to determine the efficacy of the Transmucosal Herbal Periodontal Patch (THPP) compared with placebo patch (PP) in reducing gingival inflammation at the site of placement in diabetic patients. We also aim to determine if the THPP decreases gingival inflammation throughout the mouth and the safety of THPP compared with placebo patch when applied to the mucosa in the treatment of gingival inflammation in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 85 years
* Patients must have a minimum of 3 posterior teeth in all quadrants
* A mean gingival index (GI) of >1.5 on the posterior teeth
* Diagnosis of Diabetes type 1 or 2, adequately controlled by diet and/or medications, as determined by the patient's physician

Exclusion Criteria:

* Allergy to any herbal medications
* Pregnancy or lactation
* Periodontal treatment in the last three months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08

PRIMARY OUTCOMES:
The primary endpoint of the study will be the comparison between THPP and PP in reducing the gingival index (GI) at the site of patch placement | 5 days

SECONDARY OUTCOMES:
frequency and severity of any adverse event | 5 days
Beta-glucuronidase enzyme found in gingival crevicular fluid (GCF) of the tested sites. The GCF will be collected from the second most posterior tooth in all four quadrants. | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Oded Yaniv, DMD, Principal Investigator — Izun Pharma Limited
Locations (1):
- Herzog Hospital, Jerusalem, Israel